CLINICAL TRIAL: NCT02867722
Title: Daylight Photodynamic Therapy for the Treatment of Actinic Keratoses in the Northeast United States
Acronym: DaylightPDT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI decided to not proceed with the trial due to lack of funding.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Emily Stamell Ruiz, Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000913
Record Dates: First submitted 2016-07-18; First posted 2016-08-16 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Actinic Keratosis; Non-melanoma Skin Cancer
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daylight PDT (Experimental): Patients will receive daylight-PDT treatment (aminolevulinic acid)
  Interventions: Drug: aminolevulinic acid HCl

INTERVENTIONS:
Drug: aminolevulinic acid HCl — Drug will be administered to consented patients
  Other Names: Levulan

SUMMARY:
In this study, daylight PDT will be administered to interested patients at Dana-Farber/Brigham and Women's Cancer Center. Daylight PDT has been shown to be an effective and painless alternative to traditional PDT. Daylight PDT involves application of the photosensitizer in the physician's office followed by exposure to daylight.

DETAILED DESCRIPTION:
The principal investigator will inform patients about the study during their initial consultation at the Mohs and Dermatologic Surgery Center, Dana-Farber/Brigham and Women's Cancer Center at Faulkner Hospital. The patients will be encouraged to make further inquiries about the study if they are interested. Informed consent will be obtained prior to initiating the treatment. If patients are interested in taking part in the study, the investigator will approach them in private to review the consent form and address any study-related questions.

A clinical examination along with photographs will be performed prior to application of the photosensitizer to determine the baseline number of actinic keratoses. The treatment steps were adapted from the daylight-PDT protocol presented in the phase III European multicenter study.9 The treatment will be performed if the temperature conditions are suitable to stay outdoors for 2.5 hours and not under any rainy weather conditions; however, treatment can be performed on overcast days. Suitable weather conditions include an outdoor temperature greater than 50 and between the months of April and November. This is based on a minimum of 8 J cm-2 (although other studies have shown that only 3.5 J cm-2) protoporphyrin IX light dose. A study of various geographic regions found this minimum dose was present in Turin, Italy, which is a similar latitude to Boston, MA.10 Weather conditions will be recorded on the day of treatment and final analysis will be stratified by temperature and weather conditions to evaluate whether this has impacted treatment. Subjects will be advised of the treatment requirements at the time of appointment booking and will be instructed to call the morning of their appointment to confirm that treatment can proceed. Subjects will scrub their faces with warm soapy water to clean and descale the skin and any hypertrophic AKs will be curetted. A chemical sunscreen will be applied to all sun exposed areas followed by one applicator of ALA (Levulan, DUSA pharmaceuticals, Wilmington, MA) to each treatment area. Subjects will be instructed to be exposed to daylight within 30-60 minutes of application and will remain outside in the shade for two and a half hours. Subjects will then remove the ALA and will be instructed to minimize sun exposure and to apply a physical sunscreen (zinc oxide or titanium dioxide) and wear protective clothing for the next 48 hours. This protocol will be repeated after one month unless complete response is documented at the month follow up. Subjects with a history of HSV infection will receive prophylaxis valtrex 500mg daily for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years referred for the treatment of 5 or more visible or palpable actinic keratoses on one treatment area

Exclusion Criteria:

* Age less than 18 years of age.
* Pregnant women.
* Non-English speaking patients.
* Treatment of actinic keratoses with other modalities including topical 5-fluorouracil, topical imiquimod, conventional PDT, alpha-hydroxy-acids, and glycolic acids within 2 months
* Use of retinoids within 1 month
* Use of the following medications: griseofulvin, thiazide diuretics, sulfonyureas, phenothiazines, sulfonamides, and tetracyclines
* History of cutaneous photosensitivity, lupus, porphyrias, or any other photosensitizing condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with reduction in the number of actinic keratoses after daylight PDT treatment | 1 year and 5 years

SECONDARY OUTCOMES:
Number of non-melanoma skin cancers at 1- and 5-years compared to the number of skin | 1 year and 5 years
Number of patients with treatment related adverse events as assessed by CTCAE v4.0 | 5 years
Measure patient satisfaction at 1- and 5- years using the Treatment Satisfaction Questionnaire for Medication | 1 year and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Emily Stamell Ruiz, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No
Data will be aggregated and analyzed